CLINICAL TRIAL: NCT03390231
Title: Molecular Mechanisms Underlying Stem Cell Educator Therapy for the Treatment of Diabetes
Brief Title: Stem Cell Educator Therapy in Diabetes
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Throne Biotechnologies Inc. (Industry)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2017-059-01
Record Dates: First submitted 2017-11-14; First posted 2018-01-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
Keywords: Stem Cell Educator; Immune modulation; Diabetes; Autoimmune; Insulin resistance; Pancreatic islets
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: In this project, the optimized SCE therapy for diabetes will be tested in a prospective, single-arm, open-label, single-center study
Masking Description: Open-label study with all subjects received SCE therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Stem Cell Educator (Experimental): The Stem Cell Educator (SCE) technology involves a closed-loop system that circulates a patient's blood through a blood cell separator, briefly cocultures the patient's immune cells with adherent CB-SCs in vitro, and returns only the "educated" immune cells to the patient's circulation. Several mechanistic studies with clinical samples and animal models have been conducted to demonstrate the proof of concept and clinical safety of SCE therapy. They suggest that SCE therapy may function via CB-SC induction of immune tolerance in the autoimmune T cells and pathogenic monocytes/macrophages that are encountered through the action of the autoimmune regulator (AIRE) and other molecular mechanisms. Following induction of immune tolerance in the immune cells, the immune balance and homeostasis may be restored when treated cells are returned in vivo.
  Interventions: Combination Product: Stem Cell Educator therapy

INTERVENTIONS:
Combination Product: Stem Cell Educator therapy — It briefly cocultures the patient's lymphocytes with CB-SCs in vitro, induces immune tolerance through the action of autoimmune regulator (AIRE, expressed by CB-SCs), returns the educated autologous lymphocytes to the patient's circulation, and restores immune balance and homeostasis.

SUMMARY:
Stem Cell Educator (SCE) therapy circulates a patient's blood through a blood cell separator, briefly cocultures the patient's immune cells with adherent Cord Blood Stem Cells (CB-SCs) in vitro, and returns only the "educated" autologous immune cells to the patient's circulation. Several mechanistic studies with clinical samples and animal models have demonstrated the proof of concept and clinical safety of SCE therapy. They suggest SCE therapy may function via CB-SC induction of immune tolerance in the autoimmune T cells and pathogenic monocytes/macrophages when these are exposed to the autoimmune regulator protein (AIRE) in the CB-SCs. In this project, the optimized SCE therapy for type 1 diabetes (T1D) and T2D will be tested in a prospective, single-arm, open-label, single-center study to assess its clinical efficacy and related molecular mechanisms in patients with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients are screened for enrollment in the study if both clinical signs and laboratory tests meet the diagnosis standards of American Diabetes Association.

Exclusion Criteria:

* Exclusion criteria are any clinically significant diseases in liver, kidney, and heart. Additional exclusion criteria are no pregnancy, no immunosuppressive medication, no viral diseases or diseases associated with immunodeficiency.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-27 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of inflammation-related markers in diabetic patients after Stem Cell Educator therapy | 30 days
  After treatment for 30 days, diabetic patients will be tested for inflammation-related markers (e.g.,Th1/Th2 cytokines) by flow cytometry and compare with the baseline levels.

SECONDARY OUTCOMES:
Change in insulin resistance | 30 days
  Before treatment, test for insulin sensitivity by chip analysis as baseline; After treatment, test sensitivity levels on the 1st month.
Metabolic control in HbA1C levels | 3 months
  Before treatment, test for HbA1C levels as baseline; After treatment, repeat these testing on the 3rd month. Hemoglobin A1c (HbA1c) will be reported as the changes in percentage.
Metabolic control in blood glucose levels | 3 months
  Before treatment, test for fasting glucose as baseline; After treatment, repeat these testing on the 3rd month. The blood glucose level will be measured as mMol/L.
Metabolic control in fasting C-peptide levels | 3 months
  Before treatment, test for C-peptide levels as baseline; After treatment, repeat these testing on the 3rd month. C-peptide will be measure as ng/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Zhao, MD,PhD, Study Chair — Hackensack Meridian Health; Yiming Mu, MD,PhD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Department of Endocrinology, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Yin Z, Li H, Zhang Y, Diao Y, Li Y, Chen Y, Sun X, Fisk MB, Skidgel R, Holterman M, Prabhakar B, Mazzone T. Reversal of type 1 diabetes via islet beta cell regeneration following immune modulation by cord blood-derived multipotent stem cells. BMC Med. 2012 Jan 10;10:3. doi: 10.1186/1741-7015-10-3. PMID 22233865
- [Result] Zhao Y, Jiang Z, Zhao T, Ye M, Hu C, Zhou H, Yin Z, Chen Y, Zhang Y, Wang S, Shen J, Thaker H, Jain S, Li Y, Diao Y, Chen Y, Sun X, Fisk MB, Li H. Targeting insulin resistance in type 2 diabetes via immune modulation of cord blood-derived multipotent stem cells (CB-SCs) in stem cell educator therapy: phase I/II clinical trial. BMC Med. 2013 Jul 9;11:160. doi: 10.1186/1741-7015-11-160. PMID 23837842
- [Result] Delgado E, Perez-Basterrechea M, Suarez-Alvarez B, Zhou H, Revuelta EM, Garcia-Gala JM, Perez S, Alvarez-Viejo M, Menendez E, Lopez-Larrea C, Tang R, Zhu Z, Hu W, Moss T, Guindi E, Otero J, Zhao Y. Modulation of Autoimmune T-Cell Memory by Stem Cell Educator Therapy: Phase 1/2 Clinical Trial. EBioMedicine. 2015 Nov 5;2(12):2024-36. doi: 10.1016/j.ebiom.2015.11.003. eCollection 2015 Dec. PMID 26844283
- [Result] Zhao Y, Jiang Z, Delgado E, Li H, Zhou H, Hu W, Perez-Basterrechea M, Janostakova A, Tan Q, Wang J, Mao M, Yin Z, Zhang Y, Li Y, Li Q, Zhou J, Li Y, Martinez Revuelta E, Maria Garcia-Gala J, Wang H, Perez-Lopez S, Alvarez-Viejo M, Menendez E, Moss T, Guindi E, Otero J. Platelet-Derived Mitochondria Display Embryonic Stem Cell Markers and Improve Pancreatic Islet beta-cell Function in Humans. Stem Cells Transl Med. 2017 Aug;6(8):1684-1697. doi: 10.1002/sctm.17-0078. Epub 2017 Jul 7. PMID 28685960
- See also: Tianhe Stem Cell Biotechnologies — http://www.tianhecell.com/